CLINICAL TRIAL: NCT06319547
Title: Comparing Outcome of Thoracocentesis and Pigtail Catheter Drainage in Treatment of Patients With Hepatic Hydrothorax
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ashraf Abdelkareem, Resident of Tropical medicine and gastroenterology department, Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-02-07MS
Record Dates: First submitted 2024-03-12; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Hydrothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hepatic hydrothorax (Experimental): patient with hepatic hydrothorax that develop pleural effusion either unilateral or bilateral
  Interventions: Procedure: Thoracocentasis

INTERVENTIONS:
Procedure: Thoracocentasis — patients will be submitted to diagnostic pleural fluid study, chest x-ray, liver function and blood picture
  Other Names: Pigtail Catheter drainage

SUMMARY:
Hepatic hydrothorax (HH) is a pleural effusion that develops in a patient with cirrhosis and portal hypertension in the absence of cardiopulmonary disease (Lv et al., 2018). Several factors are known to contribute to the development of effusion; the most accepted mechanism of which is the direct delivery of ascitic fluid from the peritoneal cavity to the pleural cavity by "positive" intra-abdominal pressure and a "negative" intrathoracic pressure of the pleural cavity through microscopic congenital diaphragmatic defects (Han et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the following inclusion criteria were enrolled:
* Liver cirrhosis (with or without hepatocellular carcinoma).
* Hepatic hydrothorax (bilateral or unilateral).

Exclusion Criteria:

* patients with a pleural effusion due to a condition other than HH.
* who had a diagnosis of tuberculosis pleurisy, parapneumonic effusion, inflammatory pleuritis, other neoplasms, and congestive heart failure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
percentage of empyema in patients with hepatic hydrothorax after thoracocentesis | 12 months
  Patients with hepatic hydrothorax that undergo repeated thoracocentesis will be monitored for presence of any side effects as empyema

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

REFERENCES:
- [Background] Chaaban T, Kanj N, Bou Akl I. Hepatic Hydrothorax: An Updated Review on a Challenging Disease. Lung. 2019 Aug;197(4):399-405. doi: 10.1007/s00408-019-00231-6. Epub 2019 May 25. PMID 31129701
- [Background] Gilbert CR, Shojaee S, Maldonado F, Yarmus LB, Bedawi E, Feller-Kopman D, Rahman NM, Akulian JA, Gorden JA. Pleural Interventions in the Management of Hepatic Hydrothorax. Chest. 2022 Jan;161(1):276-283. doi: 10.1016/j.chest.2021.08.043. Epub 2021 Aug 12. PMID 34390708
- [Background] Avula A, Acharya S, Anwar S, Narula N, Chalhoub M, Maroun R, Thapa S, Friedman Y. Indwelling Pleural Catheter (IPC) for the Management of Hepatic Hydrothorax: The Known and the Unknown. J Bronchology Interv Pulmonol. 2022 Jul 1;29(3):179-185. doi: 10.1097/LBR.0000000000000823. Epub 2021 Nov 10. PMID 34753862
- [Background] Liu WL, Kuo PH, Ku SC, Huang PM, Yang PC. Impact of therapeutic interventions on survival of patients with hepatic hydrothorax. J Formos Med Assoc. 2010 Aug;109(8):582-8. doi: 10.1016/S0929-6646(10)60095-2. PMID 20708509